CLINICAL TRIAL: NCT05052957
Title: Phase II Trial O6-benzylguanine(BG) and Temozolomide(TMZ) Therapy of Glioblastoma Multiforme (GBM) With Infusion of Autologous P140K MGMT+Hematopoietic Progenitors to Protect Hematopoiesis
Brief Title: hSTAR GBM (Hematopoetic Stem Cell (HPC) Rescue for GBM)
Acronym: hSTAR GBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leland Metheny (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Leland Metheny, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5320; 1U01CA236215-01 (NIH)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma Multiforme; Glioblastoma Multiforme, Adult; Supratentorial Glioblastoma; Supratentorial Gliosarcoma
MeSH Terms: conditions — Glioblastoma | interventions — O(6)-benzylguanine; Temozolomide; Filgrastim; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- stem cell mobilization after radiation therapy (Experimental): Participants at University Hospitals-Seidman Cancer Center (UH-SCC) will receive stem cell mobilization after 6 weeks of standard of care (SOC) radiotherapy. Followed by SOC chemotherapy.
  Interventions: Biological: P140K-MGMT; Drug: O6-benzylguanine; Radiation: Photon Based Radiotherapy; Drug: temozolomide; Drug: Filgrastim; Drug: carmustine

INTERVENTIONS:
Biological: P140K-MGMT — Ex Vivo Cultured P140K MGMT CD34+ Cells. The transduced cells are a biological product and production is detailed in the Cellular Therapy Lab standard operating procedures and IND 14099
Drug: O6-benzylguanine — O6BG is a low molecular-weight purine analog which selectively and irreversibly inactivates the DNA-repair enzyme, O6- alkylguanine DNA-alkyltransferase.
  Other Names: BG
Radiation: Photon Based Radiotherapy — Standard of care, photon-based radiotherapy (60Gy in 30 fractions) will be performed in both arms without concomitant TMZ between to 6 weeks post-operatively. Radiotherapy will be performed at UH-SCC.
Drug: temozolomide — Temozolomide is not directly active but undergoes rapid non-enzymatic conversion at physiologic pHto the reactive compoundMTIC. The cytotoxicity of MTIC is thought to be primarily due to alkylationof DNA. Alkylation (methylation) occurs mainly at the O6 and N7 positions of guanine
  Other Names: TMZ
Drug: Filgrastim — Filgrastim is a 175 amino acid protein manufactured by recombinant DNA technology. Endogenous filgrastim is a glycoprotein produced by monocytes, fibroblasts, and endothelial cells, which regulates the production of neutrophils within the bone marrow.
  Other Names: G-CSF,Granulocyte-Colony Stimulating Factor
Drug: carmustine — BCNU is a lipid soluble agent which has alkylating properties, plus an isocyanate metabolite which interferes with DNA and RNA synthesis.
  Other Names: BCNU,bis-chloronitrosourea

SUMMARY:
This phase II trial studies the effect of P140K MGMT hematopoietic stem cells, O6-benzylguanine, temozolomide, and carmustine in treating participants with supratentorial glioblastoma or gliosarcoma who have recently had surgery to remove most or all of the brain tumor (resected). Chemotherapy drugs, such as 6-benzylguanine, temozolomide, and carmustine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing. Placing P140K MGMT, a gene that has been created in the laboratory into bone marrow making the bone more resistant to chemotherapy, allowing intra-patient dose escalation which kills more tumor cells while allowing bone marrow to survive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, newly diagnosed, supratentorial glioblastoma or gliosarcoma who have undergone gross total tumor resection or near gross total resection (resection of >85% of enhancing tumor demonstrated by MRI) are eligible up to 35 days post-operatively. Patients with primarily infratentorial disease, or with multifocal,or leptomeningeal dissemination of disease will be excluded. In general, patients will not have > 1 cm residual measurable or evaluable disease after surgical tumor resection.
* Patient must have unmethylated MGMT
* Absence Of IDH1 or IDH2mutation on tumor tissue by a CLIA-approved immunohistochemistry or DNA sequencing test on local testing
* Patients aged 18-75 years.
* ECOG performance status 0-1or Karnofsky ≥ 70.
* No myelosuppressive chemotherapy or hematopoietic cell transplantation prior to the diagnosis of GBM and no prior chemotherapy (including Gliadel BCNU wafers) for GBM
* Life expectancy of at least 12 weeks.
* No plan for hypofractionated radiation therapy
* Adequate hematologic (absolute neutrophil count (ANC)≥ 1000/mm3, platelets ≥ 100,000/mm3, Hgb ≥ 9.5, hepatic (Bilirubin ≤ 2.0 mg/dl, AST and ALT less than or equal to 3 times institutional upper limit of normal, prothrombin time <1.2 times normal), and renal (serum creatinine ≤ 2.0 mg/dl or Creatinine Clearance ≥ 60mL/min/1.73 m2for subjects with serum creatinine levels above institutional normal). These tests will be repeated within 2 weeks of treatment with BG and TMZ, and must meet the same criteria. -Post-operative steroids are i) tapered to ≤ 8mg dexamethasone/day(or equivalent)and ii) patient has been on a stable or decreasing steroid dose for the 7 days prior to enrollment
* Patients of child-bearing potential must agree to using single barrier contraception.
* Must be willing and able to understand provide informed consent.
* Patient must have all sutures removed prior to registration
* Patient must be considered to be clinically stable.
* The subject will be identified as a candidate for an autologous transplant via an evaluation by a transplant physician per standard of care. Participants will be screened by their transplant physician and social work for a history of substance abuse per screening tool such as SIPAT. Any participant with positive screen for significant substance abuse will undergo evaluation and must have a treatment, management plan in place and must have formal review of medical team prior to initiation of transplant procedures.
* No evidence of active infection.
* Availability of 10unstained slides or FFPE sample of tumor for molecular or histopathological studies.
* Negative screening for Hepatitis B, C and HIV

Exclusion Criteria:

* Any known medical or hereditary condition associated with immunosuppression;orothermedical illness which may jeopardize patient safety.
* Known history of HIV seropositivity. This exclusion is included for two reasons. First, there is evidence of decreased marrow reserve in HIV+ patients and antiviral treatment is associated with myelosuppression. Thus, drug treatment designed to be myelosuppressive may bemore toxic in this patient population. Second, extensive laboratory culturing of the bone marrow and peripheral blood progenitor cells is required. No preclinical samples which are HIV+ have been evaluated with the gene transfer modality proposed and thus the feasibility and safety of gene transfer and selection in HIV+ samples cannot yet be advocated. Such studies are planned so as to not preclude HIV+ patients in later studies.
* Pregnant or lactating women. There is data to indicate that BCNU and TMZ is teratogenic and carcinogenic. Thus, its use in pregnant women would confer unnecessary risk to the fetus.
* Patients with symptomatic pulmonary disease and other severe co-morbid respiratory conditions, including patients with active pulmonary infection and/or pulse oximetry < 90% and a corrected DLCO < 50% of predicted. However, subjects with a corrected DLCO in the range of 50-70% should have Pulmonologyclearance prior to intervention.
* Patients with known diagnosis heart failure or cardiac insufficiency and an LVEF of < 40%. History of acute coronary event including MI within 6 months prior to study enrollment.
* Known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmiaor bradycardia.Inability to undergo repeated MRI evaluation; or allergy or intolerance of Gadolinium-containing contrast agent.
* Active illicit drug use or diagnosis of alcoholism.
* Prior diagnosis of any malignant disease with the exception of non-melanomatous skin cancer, or carcinoma in situof the cervix, bladder, prostate, or breast, unless patient has been disease-free/in remission for ≥2 years prior to date of study enrollment.
* Mental incapacity or psychiatric illness preventing informed consent.
* History of Hepatitis B or C or Hepatitis grade ≥3 are excluded due to the potential for additional hepatotixicity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants able to complete treatment | 10 years after start of study
  To evaluate and compare the feasibility of introducing and expressing P140K MGMT cDNA using a lentiviral-based provirus in autologous hematopoietic stem cells harvested from newly diagnosed IDH-1 WT GBM with unmethylated MGMT promoter using two different sequences of stem cell mobilization.
  1. What percent of patients who enter trial can complete treatment.
Incidence of adverse events | Up to 30 days post-treatment
  proportion of participants experiencing a grade 3 or higher AE/SAE
Overall Survival | Up to 15 years post-treatment
  Median overall survival in months.

SECONDARY OUTCOMES:
Myelosuppression | 5 years
  To determine what proportion of patients who receive P140K MGMT transduced CD34 cells tolerate BG and dose escalated TMZ without myelosuppression.
  We will report % of patients who suffer grade I-5 SAES related to myelosuppression.
Detection of P140K transduced BG and TMZ resistant cells | 5 years
  % of patients with detectable P-140K-MGMT
Enrichment of P140K-MGMT | 5 years
  What % of patients have enrichment of P140K-MGMT.
Tumor Response using imaging | 5 years
  Tumor response assessed via iRANO criteria
PFS using imaging | 5 years
  PFS measured from the date of initial histological diagnosis to progression (as defined above), death, last contact, or last tumor assessment before the start of further anti-tumor therapy

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie or influence the results observed from the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data.